CLINICAL TRIAL: NCT04953221
Title: A Randomized, Double-blind, Placebo-controlled, Phase II Clinical Trial to Evaluate the Effectiveness and Safety of Spray YJ001 in the Treatment of Diabetic Peripheral Neuropathic Pain.
Brief Title: The Effect of YJ001 on Diabetic Peripheral Neuropathic Pain.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: D2020155
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- M1 Test group: YJ001 for spray, topical application on the skin, drug concentration 100mg/mL, 2 times/day (interval 11-13h), 8 sprays each time, a total of 12 weeks.
  Interventions: Drug: YJ001
- M1 control group: YJ001 simulant for spray, topical application on the skin, drug concentration 100mg/mL, 2 times/day (interval 11-13h), 8 sprays each time, a total of 12 weeks.
- M2 Test group:: YJ001 for spray, topical application on the skin, drug concentration 150mg/mL, 2 times/day (interval 11-13h), 8 sprays each time, a total of 12 weeks.
  Interventions: Drug: YJ001
- M2 control group:: YJ001 simulant for spray, topical application on the skin, drug concentration 150mg/mL, 2 times/day (interval 11-13h), 8 sprays each time, a total of 12 weeks.
- M3 Test group: YJ001 for spray, topical application on the skin, drug concentration 200mg/mL, 2 times/day (interval 11-13h), 8 sprays each time, a total of 12 weeks.
  Interventions: Drug: YJ001
- M3 control group: YJ001 simulant for spray, topical application on the skin, drug concentration 200mg/mL, 2 times/day (interval 11-13h), 8 sprays each time, a total of 12 weeks.

INTERVENTIONS:
Drug: YJ001 — Skin spray
  Groups: M1 Test group; M2 Test group:; M3 Test group

SUMMARY:
In this study, a randomized, double-blind, placebo parallel-controlled design was used to evaluate the effectiveness and safety of YJ001 spray applied to local skin in patients with diabetic peripheral neuropathic pain, and to explore the best effective dose.

DETAILED DESCRIPTION:
In this study, a randomized, double-blind, placebo parallel-controlled design was used to evaluate the effectiveness and safety of YJ001 spray applied to local skin in patients with diabetic peripheral neuropathic pain, and to explore the best effective dose.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must meet all of the following criteria to be enrolled in this study.

1. The age of screening was 18-75 years old, regardless of gender;
2. Diagnosis of type 1 or type 2 diabetes for at least 1 years;
3. Diabetic peripheral neuropathic pain was diagnosed and the duration of pain was 23 months.
4. The level of glycosylated hemoglobin was less than 9%;
5. At the screening visit, according to the 11 point digital pain intensity scale (NRS), the score was greater than or equal to 4; During the 1-week lead-in period, subjects completed at least 10 NRS pain scores, and the average pain score was greater than or equal to 4.0;
6. The subjects are willing and able to comply with the study visit arrangement, treatment plan, laboratory examination and other study procedures;
7. Those who agree to participate in the trial and sign the written informed consent.

Exclusion Criteria:

- Subjects meeting any one or more of the following criteria will not be allowed to participate in this study.

1. Have known or suspected the ingredients of spray YJ001, the ingredients of YJ001 simulant, and ASA.

   Those who are allergic to aspirin, salicylic acid or yj001 (such as 5-aminosalicylic acid, sulfasalazine and salicylate) or have serious adverse reactions.
2. Those who have participated in yj001 clinical study and received research drugs.
3. The subjects have a wide range of systemic pain, which will affect the pain evaluation of the drug delivery site according to the judgment of the researchers; Or in the hand or more proximal area than the foot.
4. The subjects with severe peripheral vascular disease (such as intermittent claudication) at the time of screening were not suitable for the trial according to the judgment of the researchers.
5. Subjects suffered from nondiabetic peripheral neuropathy, such as osteoarthritis, II stage and above peripheral arterial disease, lumbar disc herniation, vitamin B deficiency, alcoholism, herpes neuralgia, vasculitis, and severe mental disorders such as depression and anxiety. It will also affect the researchers' evaluation of diabetic peripheral neuropathic pain.
6. There is skin disease in the affected skin area. According to the judgement of the researcher, it may affect the evaluation of diabetic peripheral neuropathic pain. According to the judgment of the researcher, the subjects have tattoos or other skin abnormalities that may interfere with the purpose of the study.
7. The score of skin condition evaluation of the administration site was more than 2.
8. Patients with malignant tumors, but have received appropriate treatment or resection of non metastatic skin basal cell carcinoma or squamous cell carcinoma, or cervical cancer in situ.
9. Amputation beyond the end of the fingers and toes.
10. Diabetic foot ulcers, infection and gangrene were associated with diabetes.
11. There are metabolic complications of acute diabetes, such as diabetic ketoacidosis or lactic acidosis or hyperosmolar hyperglycemia syndrome or hyperosmolar diabetic hyperglycemia.
12. One or more severe hypoglycemia events occurred 6 months before screening or during the induction period (it means that the subjects need help from others to obtain carbohydrates, glucagon or other rescue measures).
13. The NRS score of subjects with more than two pain scores was less than 3 points in the 1-week lead-in period.
14. Patients who had used transcutaneous electrical nerve stimulation (TENS), acupuncture and other treatment measures within 2 weeks before entering the group, or during the treatment period, subjects need combined transcutaneous electrical nerve stimulation (TENS) or acupuncture treatment.
15. Local analgesics (such as capsaicin patches and lidocaine patches) used in the treatment of diabetic peripheral neuropathic pain in the first 2 weeks.
16. Abnormal liver and kidney function: ast or aut > 2.5 times the upper limit of normal value, creatinine > 1.5 times the upper limit of normal value.
17. Complicated with severe cardiovascular and cerebrovascular diseases (such as degree II or III heart block, congestive heart failure with NYHA cardiac function grade III-IV, myocardial infarction, and acute stroke).
18. Severe diseases of respiratory system, blood and hematopoietic system were found.
19. There are other neurological diseases (such as cognitive impairment). The researchers believe that it may affect the evaluation of diabetic peripheral neuropathic pain or affect self ratings, or the psychiatric patients who are not suitable for the trial by the researchers.
20. Patients with known or suspected history of alcohol abuse, drug abuse or dependence in the past year.
21. Pregnant and lactating women; The male subjects (including their female partners) and the fertile female subjects had the intention of having children or could not guarantee the use of one or more contraceptives within 3 months from the beginning of screening to the end of the trial.
22. Those who participated in other clinical trials within 3 months before screening.
23. Other cases that the researcher considered unsuitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic peripheral neuropathic pain patients
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
The change in the average weekly NRS score of pain from baseline | at the twelfth week after treatment
  Numerical Rating Scale ：0-10 points, the greater the score, the more severe the pain.

SECONDARY OUTCOMES:
The change in the average weekly NRS score of pain from the baseline | 1-11 weeks after treatment
  Numerical Rating Scale ：0-10 points, the greater the score, the more severe the pain.
Changes from baseline in the average sleep disturbance scores | each week and during the follow-up period from 1 to 12 weeks after treatment
  sleep disturbance scores：0-10 points, the greater the score, the more severe the sleep disturbance.
The change from baseline in the SF-36 Quality of Life Scale score | at the 12th week after treatment
  SF-36 Quality of Life Scale score：0-100 points, the smaller the score, the more severe the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No